CLINICAL TRIAL: NCT04779424
Title: Prevalence and Incidence of Antibodies Against SARS-CoV-2 Among Primary Healthcare Providers in Belgium During One Year of the COVID-19 Epidemic
Brief Title: Prevalence and Incidence of Antibodies Against SARS-CoV-2 Among Primary Healthcare Providers in Belgium (COVID-19)
Acronym: CHARMING
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Sciensano (Other Government); University of Liege (Other)
Responsible Party: Principal Investigator, Samuel Coenen, MD PhD, Professor Clinical Epidemiology - Principal investigator, Universiteit Antwerpen
Other Study IDs: OZ8478
Record Dates: First submitted 2021-02-22; First posted 2021-03-03 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: SARS-CoV-2; COVID-19
Keywords: Seroepidemiologic Studies; Primary Health Care
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Capillary blood sample antibody point of care test
  2. Serum blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Health Care Providers (PHCPs): Any Belgian general practitioner (GP) (including those in professional training) currently working in primary care and any other primary health care providers (PHCPs) from the same GP practice who physically manage (examine, test, treat) patients/clients (frontline PHCP).
  Interventions: Other: POCT

INTERVENTIONS:
Other: POCT — Capillary blood sample antibody point of care test

SUMMARY:
This protocol focuses on the seroprevalence in primary care health care providers (PHCPs) in Belgium.

PHCPs manage the vast majority of COVID-19 and other patients and therefore are essential to organize health care efficiently. Currently however, evidence is lacking on

1. how many PHCPs get infected or diseased in Belgium,
2. the rate at which this happens,
3. their clinical spectrum,
4. their risk factors,
5. the effectiveness of the measures to prevent this from happening and
6. the accuracy of the immunological serology-based point-of-care test in a primary care setting.

This study will be set up as a prospective cohort study. All Belgian GPs in clinical practice will be invited to register online for participation in this national epidemiological study and will be asked to invite the other PHCPs in their practice to do the same. A model and demography-informed sample of registered GPs and other PHCPs will be selected. These participants will be asked at each testing point to perform a capillary blood sample antibody point of care test (OrientGene®) and complete an online questionnaire. All data analysis will be performed and reported after each relevant testing period and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Any Belgian general practitioner (GP) (including those in professional training) currently working in primary care and any other primary health care providers (PHCPs) from the same GP practice who physically manage (examine, test, treat) patients/clients (frontline PHCP), are able to comply with the study protocol and provided informed consent to participate in the study. Also PHCPs having been diagnosed with COVID-19 are included.

Exclusion Criteria:

* Staff hired on a temporary (interim) basis will be excluded as follow-up over time will be compromised.
* Administrative staff or technical staff without any contact with patients/clients will also be excluded.
* PHCPs who were not active during the inclusion period will automatically be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any Belgian general practitioner (GP) (including those in professional training) currently working in primary care and any other primary health care providers (PHCPs) from the same GP practice who physically manage (examine, test, treat) patients/clients (frontline PHCP).
Sampling Method: Non-Probability Sample
Enrollment: 3390 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of antibodies against SARS-CoV-2 in primary health care providers - T1 | 24/12/2020-08/01/2021
  The investigators will assess the prevalence of antibodies against SARS-CoV-2 in primary health care providers (PHCPs; general practitioners (GPs) and other PHCPs in their practice) in Belgium at timepoint 1 using a self-administered and self-reported serological point of care test based on a capillary blood sample (OrientGene(r)).
Prevalence of antibodies against SARS-CoV-2 in primary health care providers - T2 | 25/01/2021-31/1/2021
  The investigators will assess the prevalence of antibodies against SARS-CoV-2 in primary health care providers (PHCPs; general practitioners (GPs) and other PHCPs in their practice) in Belgium at timepoint 2 using a self-administered and self-reported serological point of care test based on a capillary blood sample (OrientGene(r)).
Prevalence of antibodies against SARS-CoV-2 in primary health care providers - T3 | 22-28/02/2021
  The investigators will assess the prevalence of antibodies against SARS-CoV-2 in primary health care providers (PHCPs; general practitioners (GPs) and other PHCPs in their practice) in Belgium at timepoint 3 using a self-administered and self-reported serological point of care test based on a capillary blood sample (OrientGene(r)).
Prevalence of antibodies against SARS-CoV-2 in primary health care providers - T4 | 22-28/03/2021
  The investigators will assess the prevalence of antibodies against SARS-CoV-2 in primary health care providers (PHCPs; general practitioners (GPs) and other PHCPs in their practice) in Belgium at timepoint 4 using a self-administered and self-reported serological point of care test based on a capillary blood sample (OrientGene(r)).
Prevalence of antibodies against SARS-CoV-2 in primary health care providers - T5 | 19-25/04/2021
  The investigators will assess the prevalence of antibodies against SARS-CoV-2 in primary health care providers (PHCPs; general practitioners (GPs) and other PHCPs in their practice) in Belgium at timepoint 5 using a self-administered and self-reported serological point of care test based on a capillary blood sample (OrientGene(r)).
Prevalence of antibodies against SARS-CoV-2 in primary health care providers - T6 | 17-23/05/2021
  The investigators will assess the prevalence of antibodies against SARS-CoV-2 in primary health care providers (PHCPs; general practitioners (GPs) and other PHCPs in their practice) in Belgium at timepoint 6 using a self-administered and self-reported serological point of care test based on a capillary blood sample (OrientGene(r)).
Prevalence of antibodies against SARS-CoV-2 in primary health care providers - T7 | 14-20/06/2021
  The investigators will assess the prevalence of antibodies against SARS-CoV-2 in primary health care providers (PHCPs; general practitioners (GPs) and other PHCPs in their practice) in Belgium at timepoint 7 using a self-administered and self-reported serological point of care test based on a capillary blood sample (OrientGene(r)).
Prevalence of antibodies against SARS-CoV-2 in primary health care providers - T8 | 13-19/09/2021
  The investigators will assess the prevalence of antibodies against SARS-CoV-2 in primary health care providers (PHCPs; general practitioners (GPs) and other PHCPs in their practice) in Belgium at timepoint 8 using a self-administered and self-reported serological point of care test based on a capillary blood sample (OrientGene(r)).
Prevalence of antibodies against SARS-CoV-2 in primary health care providers - T9 | 13-19/12/2021
  The investigators will assess the prevalence of antibodies against SARS-CoV-2 in primary health care providers (PHCPs; general practitioners (GPs) and other PHCPs in their practice) in Belgium at timepoint 9 using a self-administered and self-reported serological point of care test based on a capillary blood sample (OrientGene(r)).
Monthly incidence of antibodies against SARS-CoV-2 in primary health care providers | 24/12/2020-19/12/2021
  The investigators will assess the monthly incidence of antibodies against SARS-CoV-2 in primary health care providers (PHCPs; general practitioners (GPs) and other PHCPs in their practice) in Belgium during a 12 month follow-up period using a self-administered and self-reported serological point of care test based on a capillary blood sample (OrientGene(r)).
Annual incidence of antibodies against SARS-CoV-2 in primary health care providers | 24/12/2020-19/12/2021
  The investigators will assess the annual incidence of antibodies against SARS-CoV-2 in primary health care providers (PHCPs; general practitioners (GPs) and other PHCPs in their practice) in Belgium during a 12 month follow-up period using a self-administered and self-reported serological point of care test based on a capillary blood sample (OrientGene(r)).

SECONDARY OUTCOMES:
Longevity of antibodies against SARS-CoV-2 in primary health care providers | 24/12/2020-19/12/2021
  The investigators will assess the duration of the SARS-CoV-2 antibody response among seropositive PHCPs using a self-administered and self-reported serological point of care test based on a capillary blood sample (OrientGene(r)).
Proportion of asymptomatic cases among primary health care providers with antibodies against SARS-CoV-2 | 24/12/2020-19/12/2021
  The investigators will assess the proportion of asymptomatic cases among (new) cases (that develop during follow-up) of primary health care providers (PHCPs) with antibodies against SARS-CoV-2 based on information collected using an online questionnaire.
Determinants of of SARS-CoV-2 infection among primary health care providers | 24/12/2020-19/12/2021
  The investigators will assess the determinants of SARS-CoV-2 infection in primary health care providers (PHCPs), including PHCPs characteristics, availability and use of personal protective equipment, and exposure to COVID-19 patients, based on information collected using an online questionnaire.
Validation of a self-administered and self-reported serological point of care test in a primary care setting | 25/01/2021-31/1/2021
  The investigators will validate the immunological serology-based POCT in a primary care setting (Phase 3 validation) by assessing the sensitivity and specificity of a self-administered and self-reported serological point of care test based on capillary blood sample (OrientGene(r)) against a reference standard (laboratory serological test based on serum blood sample). As reference standard the following testing algorithm will be use, i.e. serum samples will be tested first on the ELECSYS Anti-SARS-CoV-2 S assay (Roche, Basel, Switzerland), if the cut-off index (COI) is between 0.85-3.29 the sample will be tested on the ATELLICA IM SARS-CoV-2 assay (Siemens, Munich, Germany), and if discordant results it will be tested on the LIAISON SARS-CoV-2 S1/S2 IgG assay (DiaSorin, Saluggia, Italy), using a two out of three 'reference standard'.
Familiarisation with a self-administered and self-reported serological point of care test among primary health care providers | 25/01/2021-31/1/2021
  The investigators will assess the success rate and user-friendliness of a self-administered and self-reported serological point of care test (OrientGene(r)) based on information collected using an online questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Scholtes, MD PhD, Principal Investigator — University of Liege; Elza Duysburgh, MD PhD, Principal Investigator — Sciensano
Locations (1):
- Niels Adriaenssens, Wilrijk, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. Requests can be directed at both samuel.coenen@uantwerpen.be and elza.duysburgh@sciensano.be.
Supporting Information: Study Protocol, ICF
Access Criteria: Data are available upon reasonable request. Requests can be directed at both samuel.coenen@uantwerpen.be and elza.duysburgh@sciensano.be.

REFERENCES:
- [Derived] Domen J, Abrams S, Digregorio M, Van Ngoc P, Duysburgh E, Scholtes B, Coenen S. Predictors of moderate-to-severe side-effects following COVID-19 mRNA booster vaccination: a prospective cohort study among primary health care providers in Belgium. BMC Infect Dis. 2024 Oct 10;24(1):1135. doi: 10.1186/s12879-024-09969-8. PMID 39390398
- [Derived] Domen J, Verbakel JYJ, Adriaenssens N, Scholtes B, Peeters B, Bruyndonckx R, De Sutter A, Heytens S, Van den Bruel A, Desombere I, Van Damme P, Goossens H, Buret L, Duysburgh E, Coenen S. Validation of a rapid SARS-CoV-2 antibody test in general practice. BMJ Open. 2023 May 2;13(5):e069997. doi: 10.1136/bmjopen-2022-069997. PMID 37130685
- [Derived] Adriaenssens N, Scholtes B, Bruyndonckx R, Van Ngoc P, Verbakel JYJ, De Sutter A, Heytens S, Van Den Bruel A, Desombere I, Van Damme P, Goossens H, Buret L, Duysburgh E, Coenen S. Prevalence, incidence and longevity of antibodies against SARS-CoV-2 among primary healthcare providers in Belgium: a prospective cohort study with 12 months of follow-up. BMJ Open. 2022 Sep 19;12(9):e065897. doi: 10.1136/bmjopen-2022-065897. PMID 36123069
- [Derived] Adriaenssens N, Scholtes B, Bruyndonckx R, Verbakel JY, De Sutter A, Heytens S, Van den Bruel A, Desombere I, Van Damme P, Goossens H, Buret L, Duysburgh E, Coenen S. Prevalence and incidence of antibodies against SARS-CoV-2 among primary healthcare providers in Belgium during 1 year of the COVID-19 epidemic: prospective cohort study protocol. BMJ Open. 2022 Jan 31;12(1):e054688. doi: 10.1136/bmjopen-2021-054688. PMID 35105642
- See also: link to study protocol — https://www.sciensano.be/nl/biblio/prevalence-and-incidence-antibodies-against-sars-cov-2-among-primary-healthcare-providers-belgium